CLINICAL TRIAL: NCT01570803
Title: Efficacy of Self-Expanding Nitinol S.M.A.R.T-CONTROL Stent Versus Complete SE Stent For The Atherosclerotic Femoro-Popliteal Arterial Disease : Prospective, Multicenter, Randomized, Controlled Trial (SENS-FP Trial)
Brief Title: Efficacy Between Different Two Self-Expanding Nitinol Stents For The Atherosclerotic Femoro-Popliteal Arterial Disease
Acronym: SENS-FP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study could not be initiated due to lack of research funding from the sponsors.
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Clinical Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENS-FP
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Arterial Disease; Atherosclerosis
Keywords: peripheral arterial disease,; atherosclerosis,; nitinol,; stents
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complete SE Stent (Experimental): study design is 2x2 randomization design. First, before randomization, stratification will be performed according to lesion length 15cm criteria at web-based computerized program. Patients will be randomized in a 1:1 manner according to different two (SMART versus Complete-SE) stents. And then, patients received aspirin and clopidogrel during one month. After one month from index procedure, patients were randomized to receive either clopidogrel group (clopidogrel will not be changed but continue) or cilostazol group (clopidogrel will be changed into cilostazol) in separate groups of SMART group and Complete SE group. Randomization procedure will be performed using a web-based program
  Interventions: Device: Complete SE Stent
- SMART CONTROL Stent (Active Comparator): same to Complete SE
  Interventions: Device: S.M.A.R.T CONTROL Stent

INTERVENTIONS:
Device: S.M.A.R.T CONTROL Stent — Provisional stenting should be performed; the case that optimal ballooning response is not obtained (sub-optimal balloon response) should be enrolled. The procedure is usually done, as follows; After the guidewire is passed through the target lesion, predilation of the target lesion with an optimally sized balloon will be performed prior to stent implantation. Recommended, minimal balloon dilation time is 120 seconds. The sub-optimal balloon response is defined as a residual pressure gradient of >15 mmHg, residual stenosis of >30%, and flow-limiting dissection.
  Arms: SMART CONTROL Stent
Device: Complete SE Stent — same to SMART CONTROL Stent
  Arms: Complete SE Stent

SUMMARY:
Recent stent design improvements focus on decreasing stent fracture rates which can negatively impact patency rates by rearranging strut alignment. Although there have been several retrospective or registry studies for atherosclerotic femoropopliteal disease in the East, there have been few randomized control trial for comparison of stent fracture and primary patency between different nitinol stents. Smart stent has the peak-to-valley bridge and in-line interconnection. Medtronics company have claimed Complete's stent crowns have been configured to minimize crown to crown interaction, increasing the stent's flexibility without compromising radial strength. We made the hypothesis that the design of Complete-SE stent might be more fracture-resistant or effective for in-stent restenosis, compared with Smart stent. On the other hand, 2011 ESC guideline recommended that dual antiplatelet therapy with aspirin and a thienopyridine for at least one month is recommended after infrainguinal bare-metal-stent implantation. Recent meta-analysis has shown that the efficacy of cilostazol in the atherosclerotic femoropopliteal lesion was proven. However, still specific data regarding a variety of antiplatelet regimen are limited. To date, there is no the study for comparison between clopidogrel and cilostazole in patient undergone stent implantation in femoropopliteal lesion. In conclusion, the purpose of our study is to examine and compare Primary patency and stent fracture between different two-nitinol stents (S.M.A.R.T. CONTROL versus Complete SE) and to compare binary restenosis rate between clopidogrel and cilostazol in femoropopliteal arterial lesion.

DETAILED DESCRIPTION:
Five randomized, controlled trials failed to demonstrate any benefit of a stainless-steel stent over angioplasty alone. The nitinol stent has proven superior primary patency than balloon angioplasty in superficial femoral artery (SFA) lesions. Several studies reported stent fractures were associated with a higher risk of in-stent restenosis and reocclusion. In vitro, Stefan et al. reported the 7 different SFA stents showed differences in the incidence of high strain zones, which indicates a potential for stent fracture, as demonstrated by the mechanical fatigue tests. They claimed differences in stent design might play a major role in the appearance of stent strut fracture related to restenosis and reocclusion. Also, in retrospective study, Iida et al. reported there was significant difference in stent fracture between S.M.A.R.T. stent group and Luminexx stent group and primary patency was worse in those associated with stent fracture than in those without stent fractures. Recent stent design improvements focus on decreasing stent fracture rates which can negatively impact patency rates by rearranging strut alignment.

The design of self-expandible nitinol stents might be different depending on the developed time; The first-generation nitinol stents (e.g., LuminexxTM and SmartTM) showed a remarkably high rate of stent strut fracture. A second generation of slotted tube nitinol stents has been developed. These stents had a better flexibility, by reducing the number of connections between cells or crowns, and by configurating spiral orientation of these interconnections. Several studies reported that these nitinol stents are more fracture-resistant and more flexible, some of them providing superior patency rate (e.g., LifeTM and EverflexTM). However, the one of the important limitations to their studies is that those was the non-randomized study of relative small sample size or was confined to in-vitro. Upto date, the multicenter, randomized controlled trial for direct comparison of stent fracture and primary patency between two different nitinol stents has not been done except one study; SMART versus Luminexx stent. SMART and Luminexx stent have been classified into 1st generation self-expandable nitinol stent. Complete-SE stent of Medtronic company was different to Smart stent of Cordis company in that the configuration of interconnection of Complete-SE stent had peak-to-peak connection and more spiral orientation of interconnection, compared to mart stent. On the other hand, Smart stent has the peak-to-valley bridge and in-line interconnection. Medtronics company have claimed Complete's stent crowns have been configured to minimize crown to crown interaction, increasing the stent's flexibility without compromising radial strength. We made the hypothesis that the design of Complete-SE stent might be more fracture-resistant or effective for in-stent restenosis, compared with Smart stent.

On the other hand, to date, in previous many reports, the dual antiplatelet therapy consisted of aspirin and clopidogrel have proven to decrease the incidence of cardiovascular death, myocardial infarction, or revascularization without an increase in major bleeding in patients who underwent percutaneous coronary intervention regardless of stent type (bare metal stent or drug-eluting stent). In 2011 ESC (European society of cardiology) guideline, dual antiplatelet therapy with aspirin and a thienopyridine for at least one month is recommended after infra-inguinal bare metal stent implantation (Class I, Level C). However, there have been no the definite evidence or guideline for the optimal antiplatelet agents after stent implantation one month later. There have been many studies for the efficacy of thienopyridine in peripheral arterial disease. Also, With the potential benefit of cilostazol on vascular function in vitro, there have several previous efforts to prove the efficacy of cilostazol in patients undergoing endovascular therapy or stent implantation in peripheral arterial disease. However, still specific data regarding a variety of antiplatelet regimen are limited. Also, very few trials have effectively nor properly addressed the direct comparison for the efficacy and safety between clopidogrel and cilostazol. This trial designed to evaluate the efficacy and safety between aspirin plus clopidogrel versus aspirin plus cilostazol in patients undergoing stent implantation in femoropopliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria

  1. Age 20 years of older
  2. Symptomatic peripheral-artery disease with (Rutherford 2 - 6); moderate to severe claudication (Rutherford 2-3), chronic critical limb ischemia with pain while was at rest (Rutherford 4), or with ischemic ulcers (Rutherford 5-6)
  3. Patients with signed informed consent
* Anatomical criteria

  1. Stenosis of >50% or occlusive atherosclerotic lesion of the ipsilateral femoropopliteal artery
  2. Patent (≤50% stenosis) ipsilateral iliac artery or concomitantly treatable ipsilateral iliac lesions (≤30% residual stenosis),
  3. At least one patent (less than 50% stenosed) tibioperoneal run-off vessel.

Exclusion Criteria:

1. Disagree with written informed consent
2. Major bleeding history within prior 2 months
3. Known hypersensitivity or contraindication to any of the following medication: heparin, aspirin, clopidogrel, cilostazol, or contrast agent
4. Acute limb ischemia
5. Previous bypass surgery or stenting of the ipsilateral femoropopliteal artery
6. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)
7. Patients that major amputation ("above the ankle" amputation) has been done, is planned or required
8. Patients with life expectancy <1 year due to comorbidity

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The rate of binary restenosis | one year
  the rate of binary restenosis (stenosis of at least 50 percent of the luminal diameter) or PSVR ≥ 2.5 or zero (PSVR=peak systolic velocity within the area of stenosis divided by peak systolic velocity in a normal adjacent proximal artery segment) in the treated segment at 12 months after intervention as determined by catheter angiography or Duplex ultrasound

SECONDARY OUTCOMES:
stent fracture rate, clinical outcomes, angiographic outcomes, ankle-brachial index | 1 year
  1. stent fracture rate according to fracture grade (minor, moderate, severe
  2. Limb salvage rate free of above-the-ankle amputation
  3. Sustained clinical improvement rate at 12 month follow-up
  4. Repeated target lesion revascularization (TLR) rate
  5. Repeated target extremity revascularization (TER) rate
  6. Total re-occlusion rate
  7. Comparison of angiographic variables consisted of late loss and % restenosis
  8. Ankle-brachial index (ABI) at 12 months
  9. The rate of major adverse cardiovascular events (MACE) composed of all-cause death, myocardial infarction, and stroke at 12 months
  10. Incidence of geographic miss during stent deployment due to jumping and elongation
  11. The rate of binary restenosis or PSVR ≥ 2.5 or zero according to clopidogrel and cilostazol
  12. Major bleeding rate between clopidogrel and cilostazol group.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Woon Rha, MD, PhD, Principal Investigator — Cardiovascular Center, Korea University Guro Hospital, 80, Guro-dong, Guro-gu, Seoul, 152-703, Korea
Locations (2):
- South Korea (2):
  - Cardiovascular center, Korea University Guro Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Rha SW, Choi CU, Kim EJ, Oh DJ, Cho YH, Choi WG, Lee SJ, Kim YH, Choi SH, Kim WH, Kim KC, Cho JH, Kim JH, Kim SM, Bae JH, Bong JM, Kang WY, Baek JY, Seo JB, Chung WY, Park MW, Her SH, Suh J, Kim MW, Kim YJ, Choi HJ, Soh JW; SENS-FP Investigators. Efficacy of two different self-expanding nitinol stents for atherosclerotic femoropopliteal arterial disease (SENS-FP trial): study protocol for a randomized controlled trial. Trials. 2014 Sep 10;15:355. doi: 10.1186/1745-6215-15-355. PMID 25208688